CLINICAL TRIAL: NCT02950181
Title: Descriptive Analysis of Near Infrared Spectroscopy in Critically Ill and Injured Pediatric and Neonatal Patients
Acronym: NIRSCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Concerns over standard of care and recruiting process. Investigator left UAMS, therefore study halted immediately
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202674
Record Dates: First submitted 2016-10-19; First posted 2016-11-01 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Stroke; Diabetic Ketoacidosis; Increased Intracranial Pressures; Altered Mental Status
MeSH Terms: conditions — Stroke; Diabetic Ketoacidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Specific Aim (Experimental): Correlating the NIRS/Cerebral Oximetry readings to the various critical ill and injured pediatric patients, trends, interventions, and outcomes
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Correlating the NIRS/Cerebral Oximetry readings to the various critical ill and injured pediatric patients, trends, interventions, and outcomes

SUMMARY:
This study involves looking at Cerebral oximetry measurements in pediatric and neonatal patients who are experiencing a critical illness. Such as Altered mental status, seizures, trauma, sepsis, etc.

DETAILED DESCRIPTION:
At Arkansas Children's Hospital (ACH) Pediatric Emergency Department (PED), NIRS cerebral tissue oxygenation rSO2 monitoring has become an adjunct noninvasive monitoring assessment tool along with Pulse Oximetry and End-Tidal CO2 in the critically ill and injured neonatal and pediatric patients' resuscitation endeavors or management. This has become a standard monitoring tool for patients who require medical (possible strokes, diabetic ketoacidosis, increased intracranial pressure, altered mental status, sepsis, drowning, shock, rapid sequence intubations, seizures, altered mental status, strokes, possible shunt malfunctions) or trauma (non-accidental trauma, Level One or Two Trauma with altered mental status, traumatic brain injury, altered mental status with trauma history, vascular compromise) resuscitation efforts.

Data will be collected as a retrospective and prospective chart review from the electronic medical record of patients that were treated in the pediatric emergency department of Arkansas Children's Hospital from 10-1-13 who require medical (possible strokes, diabetic ketoacidosis, increased intracranial pressure, altered mental status, sepsis, drowning, shock, rapid sequence intubations, seizures, altered mental status, strokes, possible shunt malfunctions) or trauma (non-accidental trauma, Level One or Two Trauma with altered mental status, traumatic brain injury, altered mental status with trauma history, vascular compromise) resuscitation efforts. This study will be based on the patient information recorded in these records, such as age, medications delivered, vital signs, interventions and outcomes and compared to their PED NIRS cerebral tissue oxygenation rSO2 data. All study subject materials will be assigned a unique identifying code or number. The cerebral NIRS rSO2 data will be collected/graphed and de-identified.

ELIGIBILITY:
Inclusion Criteria:

* Trauma: non-accidental trauma, Level One or Two Trauma with altered mental status, traumatic brain injury, altered mental status with trauma history, vascular compromise
* Or medical: possible strokes, diabetic ketoacidosis, increased intracranial pressure, altered mental status, sepsis, drowning, shock, rapid sequence intubations, seizures, altered mental status, strokes, possible shunt malfunctions

Exclusion Criteria:

* none

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 299 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Observing Cerebral oximetry readings when patients present to the pediatric emergency department | 4 years
  All study data will be obtained from the physical or electronic medical records obtained at Arkansas Children's Hospital. Patient's NIRS and vital signs data will be in an excel format with de-identified patient information which will be age, interventions, and etiology as denoted as Medical vs. Trauma (see study population for inclusion criteria). This is a data review with de-identified patient chart analysis for age, weight, past medical histories, co-morbidities, medical or surgical interventions, medications, seizures, duration of events, cardiac arrest, respiratory failure, intubations, and outcomes. All relevant information will be entered into a Redcap database. All study subject materials will be assigned a unique identifying code or number.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No